CLINICAL TRIAL: NCT00833651
Title: A Prospective Comparison of the Magnitude and Character of the Immune Response to Influenza Vaccine in Immunosuppressed Renal Transplant Patients and Healthy Age-matched Volunteers
Brief Title: Protective Immunity Project 02
Acronym: PIP-02
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Christian P Larsen, MD, PhD, Chairman, Dept. of Surgery, Emory University
Other Study IDs: IRB00024793; PIP-02 (Other: Other)
Record Dates: First submitted 2009-01-30; First posted 2009-02-02 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Kidney Transplant; Immunology; Immunosuppression
Keywords: Transplant; Immunology; Immunosuppression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum, PBMCs
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- tacrolimus: Recipients of primary deceased or living donor renal transplant maintained on immunosuppressive regimen utilizing tacrolimus
- sirolimus: Recipients of primary deceased or living donor renal transplant maintained on immunosuppressive regimen utilizing sirolimus
- Healthy controls: Age, gender- and race-matched individuals, not on immunosuppressive medications

SUMMARY:
Influenza (Flu) vaccine is recommended for kidney transplant patients who are at least 6 months post-transplant. The influenza vaccine stimulates the immune system to builds protective antibodies against the flu virus.

Previous research has shown that adult kidney transplant patients are not able to form as much of these protective antibodies as compared to healthy volunteers. Research has also suggested that different immunosuppressive medicines may have different effects on antibody formation. In this study, we hope to evaluate these differences in more detail.

In recent years, increasingly effective, but also increasingly complex, immunosuppressive regimens have been developed, however, there has been little detailed systematic study of the immune changes that occur in response to vaccination with these newer immunosuppressive regimens.Current policies on vaccination of transplant recipients are generic and continue to be based on old concepts rather than on any new understanding of the effects of these newer therapies on the immune system.

We hope to improve our understanding of the effects of the immunosuppressive regimens in use today (calcineurin-inhibitor, or CNI, and sirolimus-based regimens) on immune response to flu vaccine. Such knowledge will be critical to helping clinicians develop strategies for getting desirable immune responses while not causing rejection.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients between 18 and 59 years of age
2. Greater than six months post deceased or living donor renal transplant
3. Patients capable of understanding the purposes and risks of the study, who can give written informed consent and who are willing to participate in and comply with the study.
4. Patients with no known contraindications to flu vaccine (e.g. egg allergy, prior serious adverse reaction to flu vaccine, current febrile illness, marked leukopenia (WBC < 2500 cells/ml)
5. Women of childbearing potential must have a negative serum pregnancy test within 7 days of study enrollment and must not be breast-feeding.

Exclusion Criteria:

1. Patients with evidence of an active systemic infection

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Adult (ages 18-59) recipients of deceased or living donor renal transplants
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2006-11; Primary Completion 2010-02 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
To determine the effect of immunosuppressive regimens on the magnitude and character of the adaptive immune response to flu vaccine | 7, 14, 28 and 90 days post vaccination
To determine the effects of chronic immunosuppressive therapies on innate immunity during response to flu vaccine | 7, 14, 28 and 90 days post vaccination
To define the transcriptional and protein signatures of the response to flu vaccination in patients on conventional immunosuppressive regimens compared to healthy volunteers | 7, 14, 28 and 90 days post vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Christian P. Larsen, MD, DPhil, Principal Investigator — Emory University; Kenneth E Kokko, MD, PhD, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States